CLINICAL TRIAL: NCT04901299
Title: An Open-Label Phase II Trial of Fulvestrant And Neratinib in Previously Treated HRPositive, HER2-Negative Metastatic Breast Cancer Subjects Assessed With a Test Measuring Live Cell HER2 Signaling Function
Brief Title: Fulvestrant + Neratinib In Breast Cancer
Acronym: HER2-Signal
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Team decision
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Celcuity Inc (Industry); Puma Biotechnology, Inc. (Industry)
Responsible Party: Principal Investigator, Aditya Bardia, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-038
Record Dates: First submitted 2021-05-18; First posted 2021-05-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Stage IV (Metastatic) Breast Cancer; Metastatic Breast Cancer; ER Positive Breast Cancer; PR-Positive Breast Cancer; HER2-negative Breast Cancer; Invasive Breast Cancer
Keywords: stage IV (metastatic) breast cancer; Metastatic Breast Cancer; ER Positive Breast Cancer; PR-Positive Breast Cancer; HER2-negative Breast Cancer; Invasive Breast Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms | interventions — neratinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NERATINIB + FULVESTRANT (Experimental): After the screening procedures confirm participation in the research study.
  - Each Cycle = 28 days
  * Neratinib (oral, once daily)
  * Fulvestrant, injection, on 2 days for cycle 1, then one time per cycle thereafter
  Interventions: Drug: NERATINIB; Drug: FULVESTRANT

INTERVENTIONS:
Drug: NERATINIB — Neratinib will be given orally once daily on a continuous daily dosing schedule i.e., no break in dosing. Dosage per protocol
  Other Names: Nerlynx
Drug: FULVESTRANT — Fulvestrant will be given via injection every two weeks for the first 28-day cycle and every four weeks thereafter, dosage per protocol
  Other Names: Faslodex

SUMMARY:
This is a Phase 2 open label, multi-center non-randomized interventional study designed to evaluate the safety and efficacy of combining Neratinib plus Fulvestrant in previously treated metastatic HR-positive, HER2-negative breast cancer.

* This research study involves the study drug Neratinib
* The standard of care drug Fulvestrant

DETAILED DESCRIPTION:
* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

  * This research study involves the study drug Neratinib
  * The standard of care drug Fulvestrant
* It is expected that about 25 people will take part in this research study.
* This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.
* The U.S. Food and Drug Administration (FDA) has not approved Neratinib for this specific disease but it has been approved for other uses.
* The FDA has approved Fulvestrant as a treatment option for this disease. Fulvestrant is a standard of care drug that will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age).
* Histologically or cytologically confirmed stage IV (metastatic) breast cancer. PI approval is needed for patients who do not have source documentation of histologically confirmed stage IV (metastatic) breast cancer, but otherwise have known metastatic breast cancer.
* Participants must have biopsy proven HR+, i.e ER positive (ER+) and/or PR positive (PR+), HER2 non-amplified (negative), invasive breast cancer. ER, PR, and HER2 positivity would be determined per institutional (local) testing, with HR+/HER2 nonamplified (negative) status for this trial determined as per 2020 ASCO/CAP guidelines, in a biopsy/surgical specimen analyzed for ER/PR/HER2. Patients with "ER or PR low positive" (<10%) as per updated ASCO/CAP 2020 guidelines can be considered.Confirmation of adequate (15-20 unstained slides cut at 5-10 μm or 1 block) archival tissue (primary or metastatic) required before study entry. If adequate tissue not available, PI approval is required prior to study entry.
* Previously treated with no more than three prior chemotherapy regimens (no limit on prior endocrine-based regimens (including CDK4/6i and PI3K pathway inhibitors) or immunotherapy). In patients with disease recurrence during/within 12 months of (neo)adjuvant therapy, the (neo)adjuvant therapy would count as one prior regimen for this criterion. Radiation therapy or local therapy/surgery would not count as prior regimen for this criterion. Patient who discontinued chemotherapy during/after only one cycle and/or due to adverse effects without disease progression would not count the treatment/regimen as prior regimen for this criterion. Antibody drug conjugate and PARP inhibitor treatment would count as chemotherapy regimen for this criterion.
* Hyperactive HER2 signaling activity based on results from the CELsignia test (separate pre-screening test).
* Postmenopausal women with locally advanced or metastatic BC. Patients must be postmenopausal women as defined by one of the following:

  * Women > 60 years OR
  * Women ≤ 60 years, and any one of the following:

    * LH and FSH level in the postmenopausal range according to institutional standards
    * s/p post bilateral surgical oophorectomy
* Premenopausal/perimenopausal women on gonadotropin-releasing hormone agonist (to be continued during study) and estradiol level in the postmenopausal range according to institutional standards.
* ECOG performance status = 0-2
* Measurable disease as per RECIST Version 1.1.
* Ability to understand and the willingness to undergo tissue biopsy for HER2 testing (CELsignia test). Patient has signed the Informed Consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements.
* At least 2 weeks beyond treatment (chemotherapy, targeted therapy, immunotherapy, and/or radiation therapy) or major surgery and recovered from all acute toxicities prior to randomization. (adverse events from prior anti-cancer agents need to be grade 1 or lower; grade 2 alopecia or peripheral neuropathy is permitted).
* Patient has adequate bone marrow and organ function as defined by the following laboratory values at screening:

  * Absolute neutrophil count ≥ 1.5 × 109/L
  * Platelets ≥ 75 × 109/L
  * Hemoglobin ≥ 9.0 g/dL (transfusion permitted)
  * INR ≤1.5
  * GFR or creatinine clearance ≥50 mL/min (either permitted)
  * In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 x ULN. If the patient has liver metastases, ALT and AST <5 x ULN.
  * Total bilirubin ≤1.5.0 x ULN, or direct bilirubin ≤3 x ULN in patients with well documented Gilbert's Syndrome.

Exclusion Criteria:

* Participants who have received prior neratinib or any anti-HER2 therapy for metastatic disease will not be eligible. Participants who have received prior fulvestrant (or any other endocrine therapy) will be eligible. Patients with known HER2 activating mutations (either plasma and/or tissue-based genotyping) will not be eligible.
* Participants with increasing/progressive CNS metastatic disease. Patients with asymptomatic or stable CNS metastasis are eligible, provided metastasis radiologically non-progressing for at least two weeks, and patient is not actively taking steroids (more than 20 mg of prednisone or equivalent dose).
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality including any of the following:

  * History of angina pectoris, symptomatic pericarditis, coronary artery bypass graft (CABG) or myocardial infarction within 6 months prior to study entry.
  * Known LVEF <50% (by ECHO or MUGA) and/or known documented cardiomyopathy.
  * History of cardiac failure, significant/symptomatic bradycardia, Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome or any of the following:

    * Known risk to prolong the QT interval or induce Torsade's de Pointes.
    * On screening, QTcF >470 screening ECG.
* HIV-positive participants on combination antiretroviral therapy are ineligible. These participants are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Pregnant women are excluded from this study because the safety of study medications is not established in pregnant women.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, or fertile men, unless they are using highly effective methods of contraception throughout the study and after study drug discontinuation (till seven months in women and four months in males, post-study). Male patient should not donate sperm while on treatment and up to 6 months after last dose. Women are considered postmenopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential. Highly effective contraception methods include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
  * In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Note: While oral contraceptives are allowed, they should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rates (ORR) | Up to 33 Months
  ORR is defined as the proportion of patients with a confirmed CR or PR per Investigator's assessment per RECIST v1.1

SECONDARY OUTCOMES:
Time-to-Tumor Response (TTR) | Up to 33 Months
  defined for patients with confirmed objective response (CR or PR) as the time from the first dose of study treatment to the first documentation of objective tumor response
Cumulative Objective Response Incidence | Up to 33 Months
  defined as the cumulative proportion of patients with an objective response (CR or PR) after study treatment. The cumulative number of patients with an OR will be determined at the end of each time period and the cumulative incidence will then be calculated.
Duration of response (DOR) | Up to 33 Months
  is defined for patients with confirmed objective response (CR or PR) as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first. DR will be analyzed using Kaplan-Meier methods and descriptive statistics.
Progression-Free Survival (PFS) | Up to 33 Months
  defined as the time from the first dose of study treatment to the date of progression by RECIST v1.1 or death due to any cause, whichever occurs first. PFS will be analyzed using Kaplan-Meier methods and descriptive statistics.
Overall survival (OS) | Up to 33 Months
  defined as the time from the first dose of study treatment to the date of death. OS will be analyzed using Kaplan-Meier methods and descriptive statistics.
Number of Participants with Treatment Related Adverse Events as Assessed NCI CTCAE (version 5.0) | first treatment day to death up to 33 Months
  NCI CTCAE (version 5.0) criteria for adverse events
CELsignia score and Objective Response | Up to 33 Months
  The correlation between quantitative CELsignia score and OR, will be assessed to evaluate different cut-off values and corresponding treatment responses. CELsignia HER2 Pathway Activity Test
CELsignia score and CB | Up to 33 Months
  The correlation between quantitative CELsignia score and CB, will be assessed to evaluate different cut-off values and corresponding treatment responses. (CELsignia HER2 Pathway Activity Test)
CELsignia score and Progression Free Survival | up to 33 months
  The correlation between quantitative CELsignia score and PFS, will be assessed to evaluate different cut-off values and corresponding treatment responses. (CELsignia HER2 Pathway Activity Test)
CELsignia score and molecular alterations in plasma | Up to 33 Months
  The correlation between quantitative CELsignia score and molecular alterations in plasma, particularly HER2 mutations. ( CELsignia HER2 Pathway Activity Test)

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Bardia, MD,MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation